CLINICAL TRIAL: NCT00659945
Title: Efficacy of Pre-operative Aprepitant Plus Ondansetron vs Ondansetron Plus Placebo in Patients at Moderate-to-High Risk Post-operative Nausea (PONV) Undergoing Ambulatory Plastic Surgery
Brief Title: Aprepitant for PONV Prophylaxis in Outpatient Plastic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Manuel C. Vallejo, Professor, Dept. of Anesthesiology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO07070325
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Results first posted 2011-12-07 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperation, nausea, vomiting, anesthesia, plastic surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Aprepitant; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pre-op Aprepitant plus Ondansetron for PONV prophylaxis in patients undergoing outpatient plastic surgery
  Interventions: Drug: Aprepitant plus Ondansetron
- 2 (Placebo Comparator): Pre-op Placebo plus Ondansetron for PONV prophylaxis in patients undergoing outpatient plastic surgery
  Interventions: Drug: Ondansetron plus placebo

INTERVENTIONS:
Drug: Aprepitant plus Ondansetron — Aprepitant plus Ondansetron
  Other Names: Emend
  Arms: 1
Drug: Ondansetron plus placebo — Ondansetron plus placebo
  Other Names: Zofran
  Arms: 2

SUMMARY:
Hypothesis: Aprepitant plus ondansetron is more effective than ondansetron plus placebo for prevention of postoperative emesis in patients at moderate-to-high risk for PONV for up to 48 hours after surgery.

Specific Aim: To determine the incidence of PONV during the first 48 hours after surgery; in patients who have received aprepitant plus ondansetron versus ondansetron plus placebo for up to 48 hours after surgery.

DETAILED DESCRIPTION:
We plan to enroll women and men undergoing outpatient plastic surgical procedures under general anesthesia. Patients who are scheduled for outpatient plastic surgery will be contacted by one of the investigators, who would be involved in the care of the patient, as soon as they come to the hospital on the day of surgery. The patient will be given information regarding the study. After hospital registration and ample time to consider the study, the patient will be re-approached, and written informed consent will then be obtained. After informed consent is obtained, patients will be screened by one of the investigators for study eligibility.

Patients will be screened to evaluate if they are at high risk for PONV. Moderate-to-high risk for PONV includes having at least 2-3 of 5 risk factors. These five factors are: 1) female gender, 2) history of PONV, 3) history of motion sickness, 4) nonsmoking status, and 5) postoperative use of opioids. Women who report 3 of the 5 risk factors, and men who report 2 of the 5 risk factors, will be considered eligible for the study. As is the standard of care at Magee-Womens Hospital, all women of reproductive age are routinely screened for pregnancy and any patients who are pregnant will be informed and excluded from the study. Patients who are known in advance to be admitted (to either 23 hour observation or a formal hospital admission) will also be excluded from the study.

This is a prospective, randomized, double blind trial. Patients will be randomized by a computer generated number table to one of two groups (Group 1 - aprepitant, or Group 2 - placebo) within 3 hours before induction of anesthesia, consistent with the product package insert for aprepitant.

The standard of care in patients at moderate-to-high risk for PONV is to give prophylactic intravenous 5HT-3 antagonists (i.e. ondansetron). Therefore, all patients will receive PONV prophylaxis (ondansetron 4 mg intravenously) on induction of anesthesia.

All patients will receive a standardized general anesthetic which will include the following. Midazolam (2 mg) will be given intravenously for anxiolysis premedication. Medications used for induction of anesthesia will include; propofol (2-3 mg/ kg), rocuronium (0.6-0.8 mg/kg), and ondansetron (4 mg). Maintenance of general anesthesia will consist of sevoflurane (1.5 - 2.5%) in oxygen, fentanyl as needed for analgesia (not to exceed 10 μg/kg). Incremental doses of rocuronium will be used as necessary for muscle relaxation. Muscle relaxation will be reversed at the end of surgery with glycopyrrolate (0.01mg/kg) and neostigmine (0.05mg/kg). Criteria for reversal with neostigmine will be standardized in order to avoid the possibility of a repeat dose of the neostigmine, which in repeated doses is known to cause emesis.

Postoperative pain and nausea will be treated as required. If patients have PONV, all patients in both groups will receive the same rescue medications. No patient in either group will be denied rescue PONV medication. Refractory nausea and vomiting will be treated initially with an additional 4 mg dose of ondansetron (IV), then propofol (20 mg IV in divided doses), then haloperidol (2 mg IV), then dexamethasone (4 mg IV), then promethazine (6.25 mg IV, after re-verification of patency of the intravenous catheter), and metoclopramide (10 mg IV). Patients with continuing PONV refractory to these modalities will be admitted to the hospital for 23 hour observation.

Postoperative pain will be treated with fentanyl IV, and doses will be recorded. When the patient is able to tolerate oral medications, ibuprofen 400 mg PO and acetaminophen 1000 mg PO will be prescribed every 8 hours around-the-clock (i.e., regardless of reported pain scores). Immediate-release oxycodone will also be prescribed, and patients will be instructed to take 5 mg increments as frequently as every 3 hours, if needed, commensurate with verbal pain scores. If the patient reports pain scores of 5-6 out of 10, then 5 mg will be taken. If the pain score is 7-9 out of 10, then 10 mg will be taken. If the pain score is 10 out of 10, then 15 mg will be taken.

As is the standard of care at Magee-Womens Hospital, the intra-operative care, including administration of drugs will be provided by an anesthesiologist with or without the assistance of a nurse anesthetist. Nursing care in the post-anesthesia care unit (PACU) is provided by recovery room nurses, under supervision of the anesthesiologist. All drugs used in this study are approved by the Food and Drug Administration (FDA) and are routinely used at Magee-Womens Hospital for the management of patients undergoing anesthesia for surgery and treatment of PONV. The use of additional antiemetics and their dose will also be recorded for each patient. Time to discharge, delayed discharge and admission due to nausea and vomiting will be recorded.

As is the standard of care at Magee-Womens Hospital, the intra-operative care, including administration of drugs will be provided by an anesthesiologist with or without the assistance of a nurse anesthetist, or anesthesiology resident. The care in the post-anesthesia care unit (PACU) is provided by recovery room nurses, under supervision of the anesthesiologist. All drugs used in this study are approved by the Food and Drug Administration (FDA), and are routinely used at Magee-Womens Hospital for the management of patients undergoing anesthesia for the indications described herein. Time to PACU discharge eligibility (based on a score of 8 or more on the Proposed Standardized PACU Bypass/Discharge Criteria and Scoring System for Outpatients,7 time to hospital discharge eligibility (based on a score of 9 or higher on the Post-Anesthesia Discharge Score,8 and any unplanned hospital admissions (including those for PONV) will be recorded. Patients with unplanned admissions will not be excluded from further study proceedings.

Patients will be evaluated for nausea using a visual analog scale (VAS); 0 = no nausea and 10 = worst nausea ever. The presence of retching or emesis (vomiting) will be evaluated as yes or no. Nausea and vomiting will be evaluated on admission to the PACU, and at hourly intervals until discharge from the hospital. While at home; patients will be asked to fill out a structured diary to rate their nausea (0 to 10), if they retched or vomited (or not), and analgesics consumed. Patients will be asked to fill out their structured diary every four hours while awake for up to 24 hours after the first day of surgery, and every 8 hours while awake during the second day after surgery (48 hours). The information from the patient diary will be obtained by a follow-up phone interview.

This will be a randomized double blind trial. Patients will be randomized by computer program (Quattro Pro, Corel Corporation) into one of two groups, and will have a 50% chance of being in either group (Group 1 - Aprepitant or Group 2 - placebo). Both the investigator recording the observations in the PACU and the patient will be blinded to the treatment group. Data will be collected in the PACU by a blinded investigator. The patient will maintain a daily log for 48 hours and this information will be obtained by a follow-up phone interview by a blinded investigator.

Data collected from the patient's medical record will include demographic data (age, height, and weight) and these parameters will be compared using the student t test. Risk factors for PONV including (history of PONV or history of motion sickness, nonsmokers, postoperative use of opioids and female gender; descriptive statistics analysis). Other measured variables will include: incidence of nausea and emesis during the time periods described above (i.e. PACU admission and at hourly intervals until discharge, every four hours while awake for up to 24 hours after the first day of surgery, and every 8 hours while awake during the second day (48 hours) after surgery). Our primary endpoint will be the incidence of emesis at 48 hours after surgery and will be analyzed using Chi-square. Secondary endpoints will include the incidence of nausea (Mann-Whitney test) and emesis (Chi-square test) during the time periods measured above, the use and doses of rescue anti-emetics (use via Chi-square; dose via student t test), and analgesic requirements (use via Chi-squared; dose via student t test) during these time periods. Time to eligibility for PACU discharge and hospital discharged (student t test) using the aforementioned criteria will also be measured, and all unplanned hospital admissions (Chi-square) will be recorded.

A sample size of 69 patients per group is necessary to detect a significant decrease in the incidence of emesis from 33% in the placebo group to 15% in the aprepitant group using a Chi-square test assuming an alpha value of 0.05 and power of 80% (NQuery 4.0™). To allow for patients who may not complete the study, 75 patients per group (150 total patients) will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ASA (American Society of Anesthesiologists physical status) 1-3
* Male and female Age 18 to 65 years
* Plastic surgical procedure (Breast, Face, Liposuction, etc., and excluding peripheral procedures such as hand surgery and limited-scope split-thickness skin grafts) of at least 1 hour in duration
* General anesthesia
* Presence of 2 (men)/3 (women) or more risk factors for PONV
* Ambulatory surgery with same-day discharge planned

Exclusion Criteria:

* Patient refusal
* Patients who have received other antiemetics prior to their procedure
* History of allergy or sensitivity to study drugs
* Pregnancy - Patients are asked date of last menstrual period, use of birth control, tubal ligation, if they have had unprotected sexual intercourse and if they think if there is any possibility of being pregnant, and when appropriate, a pregnancy test will be obtained which is the standard of care at Magee-Womens Hospital.
* Patients with a history of chronic opioid use (chronic pain syndrome) as these patients will be less likely to have PONV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel C Vallejo, MD, Principal Investigator — Physician Services Division (UPP and CMI) | UPP | Anesthesiology and Pain Medicine
Locations (1):
- UPMC Magee Women's Hospital, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective, double blinded, randomized, two arm evaluation of 150 subjects at high risk for PONV undergoing a standardized general anesthetic with ondansetron and either aprepitant or a placebo. Recruitment period was from June 2008 through November 2009 in the preoperative holding area prior to surgery.
Pre-assignment Details: Men and women between 18 and 65 years, at high risk for PONV, undergoing ambulatory plastic surgery under general anesthesia. Exclusion criteria included patient refusal, given other anti-emetics prior to their procedure, history of allergy or sensitivity to study drugs, pregnancy, chronic opioid use, and surgery under intravenous (iv) sedation.
Groups:
- Group A(Oral Aprepitant+iv Ondansetron): oral aprepitant 40 mg plus intravenous ondansetron 4 mg
- Group B(Oral Placebo+iv Ondansetron): oral placebo plus intravenous ondansetron 4 mg IV
Period: Overall Study
Arm/Group | Group A(Oral Aprepitant+iv Ondansetron) | Group B(Oral Placebo+iv Ondansetron)
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A(Oral Aprepitant+iv Ondansetron) | Group B(Oral Placebo+iv Ondansetron) | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 75 | 150
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.7 (14.3) | 45.3 (16.3) | 44.5 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 70 | 140
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150
Emesis [Number; unit: participants] — Emesis = the reflex action of ejecting stomach contents through the mouth (definition from Bantam Medical Dictionary). The condition was patients with 2 or more major risk factors were eligible for the study. Major PONV patient-related risk factors for inclusion into the study were 1) female gender 2) history of PONV or history of motion sickness 3) non-smoking status, and 4) postoperative use of opioids.
  participants | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Having Post-operative Emesis and Nausea.
Description: Postoperative emesis was measured as present or not present (nominal data) and analyzed with Chi-square; Comparison of nausea severity was performed in two ways. In those patients who exhibited nausea VRS>0, a worst nausea score for each patient was defined as the highest nausea score recorded over the 48 hours. Mann-Whitney rank sum test was used to compare worst nausea scores. Multivariate Analysis of Variance (MANOVA) was used to determine if the mean VRS (Verbal Rating Scale) score over time was significant between the two groups.
Time Frame: 48 hours post surgery
Measure: Number; unit: participants
Arm/Group | Group A(Oral Aprepitant+iv Ondansetron) | Group B(Oral Placebo+iv Ondansetron)
Number analyzed (Participants) | 75 | 75
participants | 7 | 22
Statistical Analysis 1: Comparison: Group A(Oral Aprepitant+iv Ondansetron) vs Group B(Oral Placebo+iv Ondansetron); The primary endpoint was the incidence of emesis at any time within the first 48 hours after surgery. Power analysis showed that a sample size of 69 patients per group was necessary to detect a significant decrease in the incidence of emesis from 33% in the placebo group to 15% in the aprepitant group using a Chi-square test with an alpha value of 0.05 and power of 80%; Test type: Superiority or Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Arm/Group | Group A(Oral Aprepitant+iv Ondansetron) | Group B(Oral Placebo+iv Ondansetron)
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No